CLINICAL TRIAL: NCT03816176
Title: A Phase 2, Open-Label, Non-Comparative, Multicenter Study to Evaluate the Safety and Tolerability, Efficacy and Pharmacokinetics of Isavuconazonium Sulfate for the Treatment of Invasive Aspergillosis (IA) or Invasive Mucormycosis (IM) in Pediatric Subjects
Brief Title: A Study to Evaluate Isavuconazonium Sulfate for the Treatment of Invasive Aspergillosis (IA) or Invasive Mucormycosis (IM) in Pediatric Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9766-CL-0107; 2018-003975-36 (EudraCT Number)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Invasive Mucormycosis; Invasive Aspergillosis
Keywords: ASP9766; Cresemba; BAL8557; isavuconazonium sulfate
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isavuconazonium sulfate (Experimental): Participants received 10 milligrams/killograms (mg/kg) dose of isavuconazonium sulfate every 8 hours (± 2 hours) on days 1 and 2 for a total of 6 doses (via intravenous or oral administration at the investigator's discretion) followed by once-daily maintenance dose of 10 mg/kg for up to 84 days IA or 180 days IM or until the participant had a successful outcome as judged by the investigator, whichever occured first. The route of administration could have been changed per the investigator's discretion.
  Interventions: Drug: Isavuconazonium sulfate

INTERVENTIONS:
Drug: Isavuconazonium sulfate — Intravenous (IV) infusion
  Other Names: Cresemba
Drug: Isavuconazonium sulfate — Oral capsule
  Other Names: Cresemba

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and efficacy of isavuconazonium sulfate in pediatric participants.

DETAILED DESCRIPTION:
Treatment began on Day 1 and then participants were followed for 60 days post-last dose for safety. Treatment was administered until the participant had a successful outcome or for a maximum duration of 84 days (IA) or 180 days (IM), whichever occured first.

Participants received a loading regimen of isavuconazonium sulfate (via intravenous or oral administration at the investigator's discretion), which consisted of a dose every 8 hours (± 2 hours) on Days 1 and 2 (for a total of 6 doses), followed by once daily maintenance dosing for up to 84 days (IA) or 180 days (IM) of dosing. The first maintenance dose started 12 to 24 hours after the administration of the last loading dose. Subsequent maintenance doses were administered once daily (24 hours ± 2 hours from the previous maintenance dose). The oral formulation could only be given to participants 6 years to < 18 years of age and with a body weight of at least 12 kg. Participants who were discharged from the hospital with oral capsules for at-home administration had to return weekly for study drug accountability and to receive new oral dosing supplies. Participants who began oral administration were to complete the oral dosing acceptability assessment after ingesting their first oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with IA or IM. A positive diagnosis is defined as follows:

  * Proven, probable or possible IFI per the European Organisation for Research and Treatment of Cancer/Mycoses Study Group [EORTC/MSG], 2008 criteria Note: Subjects with "possible" IFI will be eligible for enrollment; however, diagnostic tests to confirm the invasive fungal disease as "probable" or "proven" according to the EORTC/MSG criteria should be completed within 10 calendar days after the first dose of study drug
  * Note: In addition to the criteria set for mycological criteria by the EORTC/MSG in 2008, and only for subjects with an underlying hematologic malignancy or recipients of hematopoietic stem cell transplant (HSCT) who also have clinical and radiologic features consistent with invasive fungal infection, the following are acceptable:
  * Galactomannan (GM) levels (optical density index) meeting the below criteria are acceptable mycological evidence for enrollment or upgrading the diagnosis to probable IA:
  * 1. A single value for serum or bronchoalveolar lavage (BAL) fluid of ≥ 1.0 or
  * 2. Two serum GM values of ≥ 0.5 from two separate samples
* Subject has sufficient venous access to permit intravenous administration of study drug or the ability to swallow oral capsules
* A female subject is eligible to participate if not pregnant and at least one of the following conditions applies:

  * Not a subject who is of childbearing potential, OR
  * Subject who is of childbearing potential who agrees to follow a contraceptive guidance throughout the treatment period and for at least 30 days after the final study drug administration
* Subject and subject's parent(s) or legal guardian agree that the subject will not participate in another interventional study while on treatment with the exception of oncology trials

Exclusion Criteria:

* Subject has familial short QT syndrome, is receiving medications that are known to shorten the QT interval, or has a clinically significant abnormal ECG
* Subject has evidence of hepatic dysfunction defined as any of the following:

  * Total bilirubin (TBL) ≥ 3 times the upper limit of normal (ULN)
  * Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 5 times the ULN
  * Known cirrhosis or chronic hepatic failure
* Subject has used strong cytochrome P450 (CYP3A4) inhibitors or inducers such as ketoconazole, high dose ritonavir, rifampin/rifampicin, long acting barbiturates (e.g., phenytoin), carbamazepine and St. John's Wort in the 5 days prior to the first dose of study drug
* Subject has another IFI other than possible, probably or proven IA or IM
* Subject has chronic aspergillosis, aspergilloma or allergic bronchopulmonary aspergillosis
* Subject has received mould active systemic antifungal therapy, effective against the primary IMI, for more than four days during the seven days preceding the first dose

  * Note: Prior use of prophylactic antifungal therapy is acceptable. In case of breakthrough IA while on prophylactic mould-active azole class drugs, additional documentation will be required to be submitted to the sponsor medical monitor or designee to approve subject enrollment
* Subject has known history of allergy, hypersensitivity or any serious reaction to any of the azole class antifungals, or any components of the study drug formulation
* Subject has any condition which makes the subject unsuitable for study participation
* Subject is unlikely to survive 30 days
* Subject has received investigational drug, with the exception of oncology drug trials, or trials with investigational drugs treating graft versus host disease, within 28 days or five half-lives, whichever is longer, prior to screening

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (10):
- United States (5):
  - Children's Hospital, Los Angeles, Los Angeles, California
  - University of California - Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
- Belgium (2):
  - Site BE32001, Ghent
  - Site BE32002, Leuven
- Spain (3):
  - Site ES34002, Barcelona
  - Site ES34003, Madrid
  - Site ES34001, Madrid

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Segers H, Deville JG, Muller WJ, Manzanares A, Desai A, Neely M, Bordon V, Hanisch B, Lassaletta A, Fisher BT, Autmizguine J, Groll AH, Sinnar S, Croos-Dabrera R, Engelhardt M, Jones M, Kovanda LL, Arrieta AC. Safety, outcomes, and pharmacokinetics of isavuconazole as a treatment for invasive fungal diseases in pediatric patients: a non-comparative phase 2 trial. Antimicrob Agents Chemother. 2024 Dec 5;68(12):e0048424. doi: 10.1128/aac.00484-24. Epub 2024 Nov 14. PMID 39540734
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/9766-CL-0107/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14553&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 pediatric participants diagnosed with invasive aspergillosis (IA) or invasive mucormycosis (IM) were enrolled and received isavuconazonium sulfate.
Pre-assignment Details: Male or female participant 1 year to < 18 years of age diagnosed with IA or IM. A positive diagnosis was defined as proven, probable or possible invasive fungal infection (IFI) per the European Organisation for Research and Treatment of Cancer/Mycoses Study Group [EORTC/MSG], 2008 criteria.
Groups:
- Isavuconazonium Sulfate: Participants received 10 mg/kg dose of isavuconazonium sulfate every 8 hours (± 2 hours) on days 1 and 2 for a total of 6 doses (via intravenous or oral administration at the investigator's discretion)followed by once-daily maintenance dose of 10 mg/kg for up to 84 days for IA or 180 days for IM or until the participant had a successful outcome as judged by the investigator, whichever occured first. The route of administration could have been changed per the investigator's discretion.
Period: Overall Study
Arm/Group | Isavuconazonium Sulfate
Started (31) | 31
Completed | 19
Not Completed | 12
Not completed — Miscellaneous | 5
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were enrolled and received at least one dose of study drug.
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant administered a study drug, which does not have to have a causal relationship with this treatment. It can be any unfavorable sign, symptom, or disease temporally associated with the use of a medicinal product.
  TEAE is defined as an AE observed after starting administration of the study drug through 30 days after the last dose.
Time Frame: From first dose to 30 days after the last dose (maximum 210 Days)
Population: The safety analysis set (SAF) consisted of all participant who were enrolled and received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Participants | 29

2. Primary Outcome: Percentage of Participants With All - Cause Mortality Through Day 42
Description: All - Cause Mortality Through Day 42
Time Frame: Baseline up to 42 days
Population: FAS population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants | 6.5 [0.79 to 21.42]

3. Secondary Outcome: Percentage of Participants With All - Cause Mortality
Description: EOT was defined as anytime from "day 1 to a maximum of day 180". Data reported in the table below for each category, i.e., Day 84 represented data between Day 1 and Day 84 and for EOT, data represented between Day 1 to the EOT day for each individual. Participants who died after EOT assessment but before reaching Day 84 were included in the data for Day 84 category. Only those deaths that occurred after Day 84 would be included in EOT category if the death occurred during the treatment period (i.e. prior to the EOT).
Time Frame: Baseline up to day 84 and end of treatment (EOT) (up to a maximum of 180 days) (Average duration of treatment: 57.7 days)
Population: FAS population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 84 | 9.7 [2.04 to 25.75]
  EOT | 0.00 [0.00 to 0.00]

4. Secondary Outcome: Percentage of Participants With Overall Response: Adjudication Committee (AC) Assessment
Description: Overall response was based on a composite of clinical, mycological, and radiological responses with success criteria assessed. Success criteria as assessed by AC in:
  Clinical response:
  * Complete: Resolution of all attributable clinical symptoms and physical findings
  * Partial: Resolution of at Least some of the clinical symptoms and physical findings associated with IFD
  Mycological response:
  * Eradication: No growth of the original (at baseline) causative organism on culture or identified by histology/cytology on post baseline (after day 7) cultures and/or histology/cytology
  * Presumed eradication: Missing post baseline documentation of eradication of the original causative organism at baseline PLUS resolution of all or some clinical symptoms/physical finding
  Radiological response:
  * Complete: ≥ 90% improvement
  * Partial: At least < 25% response at day 42 and at least 50% by Day 84
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: FAS population
Measure: Number; unit: Percentage of partticipants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of partticipants
  Day 42 | 29.0
  Day 84 | 25.8
  EOT | 54.8

5. Secondary Outcome: Percentage of Participants With Clinical Response: AC Assessment
Description: AC Assessed Clinical response was defined as follows:
  * Success: Complete (if resolution of all attributable clinical symptoms and physical findings occurs); Partial (if resolution of at least some of the clinical symptoms and physical findings associated with IFD)
  * Failure: Stable (if minor of no change in clinical symptoms and physical findings associated with IFD); Progression (if worsening or new clinical symptoms and physical findings associated with IFD, or if alternative systemic antifungal treatment is required)
  * Not Evaluable: If not assessed or no clinical signs or symptoms at baseline
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: FAS population. If participant did not reach Day 42 or Day 84 of therapy then the AC did not perform these assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 42 Success | 0
  Day 42 Failure | 0
  Day 42 Not Evaluable | 58.06
  Day 42 No Assessment | 41.94
  Day 84 Success | 0
  Day 84 Failure | 0
  Day 84 Not Evaluable | 35.48
  Day 84 No Assessment | 64.52
  EOT Success | 6.45
  EOT Failure | 9.68
  EOT Not Evaluable | 83.87
  EOT No Assessment | 0

6. Secondary Outcome: Percentage of Participants With Clinical Response: Investigator Assessment
Description: Investigator-assessed Clinical Response was defined as follows:
  * Success: if resolution of all attributable signs and symptoms or resolution of attributable clinical symptoms and physical findings
  * Failure: if no resolution of any attributable signs and symptoms or no resolution of any attributable signs and symptoms (no change) or worsening of any attributable signs and symptoms
  * Not Evaluable: if results not available /participant unevaluable or if no attributable signs and symptoms
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: FAS population. If participant did not reach Day 42 or Day 84 of therapy then the investigator did not perform these assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 42 Success | 41.9
  Day 42 Failure | 9.7
  Day 42 Not Evaluable | 0
  Day 42 No Assessment | 48.4
  Day 84 Success | 32.3
  Day 84 Failure | 0
  Day 84 Not Evaluable | 0
  Day 84 No Assessment | 67.7
  EOT Success | 61.3
  EOT Failure | 29.0
  EOT Not Evaluable | 3.2
  EOT No Assessment | 6.5

7. Secondary Outcome: Percentage of Participants With Radiological Response: AC Assessment
Description: AC-assessed Radiological Response was defined as follows:
  * Success: Complete (if ≥ 90% improvement); Partial (if at least < 25% response at day 42 and at least 50% response by Day 84)
  * Failure: Stable (if minor or no change in radiographic abnormalities associated with IFD, but no signs of progression); Progression (if worsening or new radiological abnormalities associated with IRD)
  * Not Evaluable: if no post baseline radiology available with baseline evidence of radiolical disease Or Radiology not applicable at baseline
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: FAS population. If participant did not reach Day 42 or Day 84 of therapy then the AC did not perform these assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 42 Success | 29.03
  Day 42 Failure | 6.45
  Day 42 Not Evaluable | 22.58
  Day 42 No Assessment | 41.94
  Day 84 Success | 25.81
  Day 84 Failure | 0
  Day 84 Not Evaluable | 9.68
  Day 84 No Assessment | 64.52
  EOT Success | 51.61
  EOT Failure | 16.13
  EOT Not Evaluable | 32.26
  EOT No Assessment | 0

8. Secondary Outcome: Percentage of Participants With Radiological Response: Investigator Assessment
Description: Investigator's assessed radiological response was defined as follows:
  * Success: if ≥ 90% improvement, ≥ 50% to < 90% improvement, ≥ 25% to 50% improvement (for Day 42 only)
  * Failure if < 25% improvement at any time or no signs or radiological Images
  * Not Evaluable if results not evaluable or no radiological data available
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 42 Success | 25.8
  Day 42 Failure | 3.2
  Day 42 Not Evaluable | 12.9
  Day 42 No Assessment | 58.1
  Day 84 Success | 19.4
  Day 84 Failure | 0
  Day 84 Not Evaluable | 9.7
  Day 84 No Assessment | 71.0
  EOT Success | 48.4
  EOT Failure | 16.1
  EOT Not Evaluable | 29.0
  EOT No Assessment | 6.5

9. Secondary Outcome: Percentage of Participants With Mycological Response: AC Assessment
Description: AC assessed mycological response was defined as follows:
  * Success: Eradicated (no growth of the original [at baseline] causative organism on culture or identified by histology/cytology on post baseline [after day 7] cultures and/or histology/cytology); Presumed Eradicated (missing post baseline documentation of eradication of the original causative organism at baseline PLUS resolution of all or some clinical symptoms/physical finding)
  * Failure: Persistence (persistence of the original causative organism cultured or identified by histological /cytology at baseline); Presumed Persistence (missing post baseline documentation of the persistence of the original causative organism at baseline PLUS no resolution or worsening of any clinical symptoms/physical findings)
  * Not Evaluable - no mycological evidence
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: FAS population. If participant did not reach Day 42 or Day 84 of therapy then the AC did not perform these assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of participants
  Day 42 Success | 19.35
  Day 42 Failure | 3.23
  Day 42 Not Evaluable | 35.48
  Day 42 No Assessment | 41.94
  Day 84 Success | 19.35
  Day 84 Failure | 0
  Day 84 Not Evaluable | 16.13
  Day 84 No Assessment | 64.52
  EOT Success | 35.48
  EOT Failure | 12.90
  EOT Not Evaluable | 51.61
  EOT No Assessment | 0

10. Secondary Outcome: Percentage of Participats With Mycological Response: Investigator Assessment
Description: Investigator's assessed mycological response was defined as follows:
  * Success: Eradicated (no growth of the original [at baseline] causative organism on culture or identified by histology/cytology on post baseline [after day 7] cultures and/or histology/cytology); Presumed Eradicated (missing post baseline documentation of eradication of the original causative organism at baseline PLUS resolution of all or some clinical symptoms/physical finding)
  * Failure: Persistence (persistence of the original causative organism cultured or identified by histological /cytology at baseline); Presumed Persistence (missing post baseline documentation of the persistence of the original causative organism at baseline PLUS no resolution or worsening of any clinical symptoms/physical findings)
  * Not Evaluable: Indeterminate/no mycological follow-up or results available
  * No assessment: Those participants that do not fall under any of the above criteria
Time Frame: Baseline up to days 42, 84 and EOT (180 days)
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 31
Percentage of Participants
  Day 42 Success | 22.6
  Day 42 Failure | 6.5
  Day 42 Not Evaluable | 22.6
  Day 42 No Assessment | 48.4
  Day 84 Success | 25.8
  Day 84 Failure | 0
  Day 84 Not Evaluable | 3.2
  Day 84 No Assessment | 71.0
  EOT Success | 45.2
  EOT Failure | 12.9
  EOT Not Evaluable | 35.5
  EOT No Assessment | 6.5

11. Secondary Outcome: Pharmacokinetics of Isavuconazonium Sulphate in Plasma: Trough Concentration (Ctrough)
Description: Ctrough was defined as the predose concentration at the end of dosing interval.
Time Frame: Predose on days 7, and 14
Population: The pharmacokinetic analysis set (PKAS) consisted of all participants who took at least one dose of study drug and who had at least one plasma concentration.
Measure: Mean (Standard Deviation); unit: Nanograms/milliter (ng/mL)
Arm/Group | Isavuconazonium Sulfate
Number analyzed (Participants) | 28
Nanograms/milliter (ng/mL)
  Age group 1 to <6 Day 7: number analyzed (Participants) | 6
  Age group 1 to <6 Day 7 | 2965.0 (1770.5)
  Age group 1 to <6 Day 14: number analyzed (Participants) | 6
  Age group 1 to <6 Day 14 | 2286.7 (1991.3)
  Age group 6 to <12 Day 7: number analyzed (Participants) | 10
  Age group 6 to <12 Day 7 | 3732.7 (1855.0)
  Age group 6 to <12 Day 14: number analyzed (Participants) | 6
  Age group 6 to <12 Day 14 | 3623.3 (1878.0)
  Age group 12 to <18 Day 7: number analyzed (Participants) | 9
  Age group 12 to <18 Day 7 | 3862.2 (1427.1)
  Age group 12 to <18 Day 14: number analyzed (Participants) | 6
  Age group 12 to <18 Day 14 | 4380.0 (2022.4)

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after the last dose (maximum 210 days)
Description: SAF popuation
Arm/Group | Isavuconazonium Sulfate
All-Cause Mortality (participants affected / at risk) | 3/31
Serious Adverse Events (participants affected / at risk) | 18/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isavuconazonium Sulfate (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (4)
Infusion site pain (General disorders) | 1 (1)
Infusion site pruritus (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 3 (4)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Social problem (Social circumstances) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isavuconazonium Sulfate (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 (6)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Nausea (Gastrointestinal disorders) | 4 (8)
Stomatitis (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 7 (14)
Chills (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 5 (5)
Pain (General disorders) | 2 (3)
Pyrexia (General disorders) | 9 (13)
Drug hypersensitivity (Immune system disorders) | 2 (3)
COVID-19 (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 3 (4)
QRS axis abnormal (Investigations) | 2 (4)
Transaminases increased (Investigations) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Headache (Nervous system disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Pallor (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03816176/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03816176/SAP_003.pdf